CLINICAL TRIAL: NCT06846515
Title: A Phase 3 Randomized, Double-blind, Multi-center, Placebo-controlled Study to Evaluate the Efficacy and Safety of AR882 in Participants With Gout
Brief Title: Phase 3 Evaluation of Efficacy and Safety of AR882 in Gout Patients (AR882-301)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Arthrosi Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AR882-301
Record Dates: First submitted 2025-02-21; First posted 2025-02-26 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Gout; Arthritis, Gouty; Hyperuricemia; Gout Chronic
MeSH Terms: conditions — Gout; Arthritis, Gouty; Hyperuricemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- AR882 50 mg (Experimental): AR882 50 mg taken once daily for 12 months
  Interventions: Drug: AR882 50 mg
- AR882 75 mg (Experimental): AR882 75 mg taken once daily for 12 months
  Interventions: Drug: AR882 75 mg
- Placebo (Placebo Comparator): AR882 matching placebo taken once daily for 12 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AR882 50 mg — Solid Oral Capsule
  Arms: AR882 50 mg
Drug: AR882 75 mg — Solid Oral Capsule
  Arms: AR882 75 mg
Drug: Placebo — Matching Solid Oral Capsule Placebo
  Arms: Placebo

SUMMARY:
This study will assess the serum uric acid lowering effect and safety of AR882 in gout patients at two doses compared to placebo over 12 months

ELIGIBILITY:
Inclusion Criteria:

* History of gout
* Occurrence of ≥ 2 self-reported gout flares in the last 12 months
* Body weight no less than 50 kg
* Patients who are NOT on approved urate-lowering therapy (ULT) must have sUA ≥ 7 mg/dL
* Patients who are on medically appropriate ULT must have sUA > 6 mg/dL
* Serum creatinine must be < 3.0 mg/dL and estimated CLcr ≥ 30 mL/min

Exclusion Criteria:

* Malignancy within 5 years, except for successfully treated basal or squamous cell carcinoma of the skin
* Pregnant or breastfeeding
* History of symptomatic kidney stones within the past 6 months

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2025-03-11 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Serum urate (uric acid) (sUA) level < 6 mg/dL at month 6 | 24 weeks
  Comparison of the treatment groups for the proportion of patients with serum urate (uric acid) (sUA) level < 6 mg/dL at month 6

SECONDARY OUTCOMES:
Change in tophus burden by month 12 | 48 weeks
  Comparison of the treatment groups for the proportion of patients who experience a complete response, marked or partial response, of at least 1 target tophus at Month 12, with no evidence of disease progression (no new tophus or single tophus showing progression) and patients with no new tophi formation at month 12 as determined using the computer-assisted photographic evaluation in rheumatology (CAPER) method
Serum urate (uric acid) (sUA) level < 6 mg/dL from the end of month 9 to the end of month 12 | 12 weeks
  Comparison of the treatment groups for the proportion of patients with serum urate (uric acid) (sUA) level < 6 mg/dL for the 3-month period from the end of month 9 to the end of month 12
No gout flares from the end of month 9 to the end of month 12 | 12 weeks
  Comparison of the treatment groups for the proportion of patients with no gout flares for the 3-month period from the end of month 9 to the end of month 12
Incidence of Adverse Events | 56 weeks
  Treatment Emergent Adverse Events and Serious Adverse Event incidence

CONTACTS AND LOCATIONS:
Overall Officials: Robert Keenan, MD, Study Director — Arthrosi Therapeutics, Inc.
Locations (89):
- United States (89):
  - Arthrosi Investigative Site (620), Birmingham, Alabama
  - Arthrosi Investigative Site (616), Huntsville, Alabama
  - Arthrosi Investigative Site (680), Peoria, Arizona
  - Arthrosi Investigative Site (640), Phoenix, Arizona
  - Arthrosi Investigative Site (617), Little Rock, Arkansas
  - Arthrosi Investigative Site (614), Garden Grove, California
  - Arthrosi Investigative Site (618), La Mesa, California
  - Arthrosi Investigative Site (687), La Mesa, California
  - Arthrosi Investigative Site (655), La Palma, California
  - Arthrosi Investigative Site (632), Lincoln, California
  - Arthrosi Investigative Site (605), Lomita, California
  - Arthrosi Investigative Site (675), Long Beach, California
  - Arthrosi Investigative Site (603), Santa Monica, California
  - Arthrosi Investigative Site (672), Tarzana, California
  - Arthrosi Investigative Site (656), Thousand Oaks, California
  - Arthrosi Investigative Site (660), Aurora, Colorado
  - Arthrosi Investigative Site (669), Colorado Springs, Colorado
  - Arthrosi Investigative Site (612), Fort Collins, Colorado
  - Arthrosi Investigative Site (665), Cooper City, Florida
  - Arthrosi Investigative Site (613), Jupiter, Florida
  - Arthrosi Investigative Site (611), Miami, Florida
  - Arthrosi Investigative Site (644), Miami, Florida
  - Arthrosi Investigative Site (694), Palmetto Bay, Florida
  - Arthrosi Investigative Site (615), Sanford, Florida
  - Arthrosi Investigative Site (600), Tampa, Florida
  - Arthrosi Investigative Site (673), Atlanta, Georgia
  - Arthrosi Investigative Site (682), Lilburn, Georgia
  - Arthrosi Investigative Site (652), Marietta, Georgia
  - Arthrosi Investigative Site (658), Honolulu, Hawaii
  - Arthrosi Investigative Site (676), Boise, Idaho
  - Arthrosi Investigative Site (634), Meridian, Idaho
  - Arthrosi Investigative Site (657), Chicago, Illinois
  - Arthrosi Investigative Site (648), Melrose Park, Illinois
  - Arthrosi Investigative Site (678), Indianapolis, Indiana
  - Arthrosi Investigative Site (679), Overland Park, Kansas
  - Arthrosi Investigative Site (674), Louisville, Kentucky
  - Arthrosi Investigative Site (627), Mandeville, Louisiana
  - Arthrosi Investigative Site (650), New Orleans, Louisiana
  - Arthrosi Investigative Site (641), Prairieville, Louisiana
  - Arthrosi Investigative Site (662), Oxon Hill, Maryland
  - Arthrosi Investigative Site (653), Rockville, Maryland
  - Arthrosi Investigative Site (636), Fall River, Massachusetts
  - Arthrosi Investigative Site (622), Bay City, Michigan
  - Arthrosi Investigative Site (628), Farmington Hills, Michigan
  - Arthrosi Investigative Site (645), Southfield, Michigan
  - Arthrosi Investigative Site (633), Gulfport, Mississippi
  - Arthrosi Investigative Site (635), Jackson, Mississippi
  - Arthrosi Investigative Site (693), Olive Branch, Mississippi
  - Arthrosi Investigative Site (637), Springfield, Missouri
  - Arthrosi Investigative Site (626), Town and Country, Missouri
  - Arthrosi Investigative Site (664), Missoula, Montana
  - Arthrosi Investigative Site (610), Lincoln, Nebraska
  - Arthrosi Investigative Site (684), Omaha, Nebraska
  - Arthrosi Investigative Site (651), Omaha, Nebraska
  - Arthrosi Investigative Site (686), Las Vegas, Nevada
  - Arthrosi Investigative Site (661), Brooklyn, New York
  - Arthrosi Investigative Site (663), Hartsdale, New York
  - Arthrosi Investigative Site (625), Charlotte, North Carolina
  - Arthrosi Investigative Site (681), Charlotte, North Carolina
  - Arthrosi Investigative Site (683), Raleigh, North Carolina
  - Arthrosi Investigative Site (649), Shelby, North Carolina
  - Arthrosi Investigative Site (666), Fargo, North Dakota
  - Arthrosi Investigative Site (671), Mason, Ohio
  - Arthrosi Investigative Site (631), Norman, Oklahoma
  - Arthrosi Investigative Site (642), Tulsa, Oklahoma
  - Arthrosi Investigative Site (647), Horsham, Pennsylvania
  - Arthrosi Investigative Site (623), Philadelphia, Pennsylvania
  - Arthrosi Investigative Site (638), Charleston, South Carolina
  - Arthrosi Investigative Site (604), Fort Mill, South Carolina
  - Arthrosi Investigative Site (608), North Charleston, South Carolina
  - Arthrosi Investigative Site (619), Chattanooga, Tennessee
  - Arthrosi Investigative Site (624), Hendersonville, Tennessee
  - Arthrosi Investigative Site (670), Amarillo, Texas
  - Arthrosi Investigative Site (677), Austin, Texas
  - Arthrosi Investigative Site (690), Dallas, Texas
  - Arthrosi Investigative Site (639), DeSoto, Texas
  - Arthrosi Investigative Site (601), Houston, Texas
  - Arthrosi Investigative Site (688), Plano, Texas
  - Arthrosi Investigative Site (689), Prosper, Texas
  - Arthrosi Investigative Site (607), Sugar Land, Texas
  - Arthrosi Investigative Site (646), Tomball, Texas
  - Arthrosi Investigative Site (659), Tomball, Texas
  - Arthrosi Investigative Site (643), Clinton, Utah
  - Arthrosi Investigative Site (609), Salt Lake City, Utah
  - Arthrosi Investigative Site (654), Salt Lake City, Utah
  - Arthrosi Investigative Site (606), Charlottesville, Virginia
  - Arthrosi Investigative Site (691), Winchester, Virginia
  - Arthrosi Investigative Site (685), Bellevue, Washington
  - Arthrosi Investigative Site (668), Kenosha, Wisconsin

IPD SHARING:
Plan to Share IPD: No